CLINICAL TRIAL: NCT02089997
Title: Benet 75 mg Tablets Special Drug Use Surveillance: Long-term Use (12-month Treatment Survey)
Brief Title: Special Drug Use Surveillance on Long-term Use of Sodium Risedronate Tablets (Benet 75 mg Tablets) (12-month Treatment Survey)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 178-001; JapicCTI-142463 (Registry Identifier: JapicCTI); JapicCTI-R171017 (Other: JapicCTI)
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-02

CONDITIONS: Osteoporosis
Keywords: Pharmacological therapy
MeSH Terms: conditions — Osteoporosis | interventions — Risedronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 75 mg of sodium risedronate: 75 mg of sodium risedronate is administered orally with a sufficient volume (approximately 180 mL) of water once monthly after waking.
  Interventions: Drug: Sodium Risedronate

INTERVENTIONS:
Drug: Sodium Risedronate — Sodium risedronate tablets
  Other Names: Benet 75mg Tablets

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of sodium risedronate tablets (Benet 75 mg Tablets) in osteoporosis patients in daily medical practice, as well as to examine "the status of treatment compliance" - i.e., whether sodium risedronate tablets are taken properly in accordance with the prescribed once-monthly regimen

DETAILED DESCRIPTION:
This surveillance was designed to evaluate the safety and efficacy of sodium risedronate tablets (Benet 75 mg Tablets) as well as to evaluate the status of treatment compliance in osteoporosis patients in daily medical practice.

The usual dosage for adult is 75 mg of sodium risedronate administered orally with a sufficient volume (approximately 180 mL) of water once monthly after waking. For at least 30 minutes after administration, patients should avoid lying in a supine position and should avoid taking food, drink (except for water) or other oral drugs. For more details, see the "Precautions related to dosage and administration" section of the package insert.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis patients

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 3304 (Actual)
Dates: Start 2013-05-27 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 606 investigative sites in Japan from 27-May 2013 to 30-April 2016 .
Pre-assignment Details: Participants with a historical diagnosis of osteoporosis were enrolled to receive sodium risedronate 75 milligram (mg) for up to 12 months as per routine medical practice.
Groups:
- Sodium Risedronate 75 mg: Sodium risedronate 75 mg, tablet, orally, once monthly for up to 12 months.
Period: Overall Study
Arm/Group | Sodium Risedronate 75 mg
Started | 3304
Completed | 3058
Not Completed | 246
Not completed — Case report forms uncollected | 99
Not completed — Protocol Violation | 147

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set was defined as all participants who were enrolled and completed the study.
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 3058
Age, Customized [Number; unit: Participants]
  < 65 years | 373
  ≥ 65 years | 2678
  Unknown | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2817
  Male | 241
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 3058
Pregnancy Status [Number; unit: Participants] — This baseline characteristic was analyzed only in female participants.
  Participants
    Pregnant | 0
    Not pregnant | 2329
    Unknown | 488
Weight [Number; unit: Participants]
  < 50.0 kg | 1050
  ≥ 50.0 kg | 953
  Unknown | 1055
BMI [Number; unit: Participants] — Body Mass Index = weight (kg)/[height (m)^2]
  Participants
    < 18.5kg/m^2 | 162
    ≥ 18.5kg/m^2 < 25.0kg/m^2 | 1108
    ≥ 25.0kg/m^2 | 291
    Unknown | 1497
Osteoporosis Class [Number; unit: Participants]
  Primary Osteoporosis | 2696
  Secondary Osteoporosis | 232
  Unknown | 130
Predisposition to Hypersensitivity [Number; unit: Participants]
  Had No Predisposition to Hypersensitivity | 2658
  Had Predisposition to Hypersensitivity | 151
  Unknown | 249
Medical Complications [Number; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Participants may be represented in more than 1 category.
  Participants
    Had Presence of Medical Complications | 2649
    Had No Presence of Medical Complications | 409
Medical History（not Inclusive of a History of Fractures） [Number; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history and Bone Fractures were out of scope for Medical history in this study. Other medical history included all medical history except for those mentioned above. Participants may be represented in more than 1 category.
  Participants
    Had Medical History | 587
    Had No Medical History | 2264
    Unknown | 207
Pretreatment Osteoporosis Drug [Number; unit: Participants]
  Had Treatment Drug | 1149
  Had No Treatment Drug | 1909
Concomitant Medication [Number; unit: Participants]
  Had Concomitant Medication | 2512
  Had No Concomitant Medication | 546

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs)
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with administration of sodium risedronate, whether or not it was considered related to the treatment.
Time Frame: Up to Month 12
Population: Safety Analysis Set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 3058
Participants | 231

2. Secondary Outcome: Percent Change From Baseline in Mean Lumbar Spine (L2-L4) Bone Mineral Density (BMD) at Final Assessment
Description: BMD was measured with Dual-energy X-ray Absorptiometry. Reporting data are the change in BMD in the second to the fourth lumbar vertebrae, L2 to L4, and the averages of L2 to L4 at end of study relative to baseline.
Time Frame: Baseline and final assessment (up to Month 12)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 545
Percent change | 4.700 (12.118)

3. Secondary Outcome: Percent Change From Baseline in Femur (Neck Region) BMD at Final Assessment
Description: BMD was measured with Dual-energy X-ray Absorptiometry. Reporting data are the change in BMD in the femur (neck region) at end of study relative to baseline.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 393
Percent change | 1.008 (5.473)

4. Secondary Outcome: Percent Change From Baseline in Femur (Total Proximal Femur) BMD at Final Assessment
Description: BMD was measured with Dual-energy X-ray Absorptiometry. Reporting data are the change in BMD in the total proximal femur (whole bone, trochanteric region, and neck region) at end of study relative to baseline.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 424
Percent change | 1.745 (5.180)

5. Secondary Outcome: Percent Change From Baseline in Radius BMD at Final Assessment
Description: BMD was measured with Dual-energy X-ray Absorptiometry. Reporting data are the change in BMD in the radius at end of study relative to baseline.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 569
Percent change | 1.173 (6.909)

6. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Type 1 Collagen Cross-linked N-telopeptide (NTX) at Final Assessment
Description: Blood samples for serum bone turnover markers were collected at specified visits according to the study schedule.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 174
Percent change | -14.024 (27.863)

7. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Tartrate-resistant Acid Phosphatase 5b (TRACP-5b) at Final Assessment
Description: Blood samples for serum bone turnover markers were collected at specified visits according to the study schedule.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 449
Percent change | -32.016 (30.219)

8. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Bone-type Alkaline Phosphatase (BAP) at Final Assessment
Description: Blood samples for serum bone turnover markers were collected at specified visits according to the study schedule.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 128
Percent change | -19.449 (28.058)

9. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Serum Procollagen 1 N-terminal Peptide (P1NP) at Final Assessment
Description: Blood samples for serum bone turnover markers were collected at specified visits according to the study schedule.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 217
Percent change | -46.302 (30.482)

10. Secondary Outcome: Percent Change From Baseline in Bone Metabolism Markers Urinary Type 1 Collagen Cross-linked N-telopeptide (NTX) at Final Assessment
Description: Urine samples for urinary bone turnover markers were collected at specified visits according to the study schedule.
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 194
Percent change | -22.010 (60.634)

11. Secondary Outcome: Change From Baseline in Height
Time Frame: Baseline and final assessment (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 806
Centimeter | -0.37 (1.10)

12. Secondary Outcome: Number of Participants Who Had Lumbar Backache at Final Assessment
Time Frame: Final assessment (Month 12)
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Sodium Risedronate 75 mg
Number analyzed (Participants) | 2052
Participants | 663

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only ADRs were collected in this study. Participants may be represented in more than 1 category.
Arm/Group | Sodium Risedronate 75 mg
Serious Adverse Events (participants affected / at risk) | 15/3058
Other Adverse Events (participants affected / at risk) | 71/3058
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Risedronate 75 mg (N=3058)
Pneumonia (Infections and infestations) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cardiac hypertrophy (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Collagen disorder (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Death (General disorders) | 2 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sodium Risedronate 75 mg (N=3058)
Diarrhoea (Gastrointestinal disorders) | 19
Nausea (Gastrointestinal disorders) | 28
Pyrexia (General disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.